CLINICAL TRIAL: NCT05162144
Title: Proximal Medial Gastriocnemius Recession for Chronic Plantar Fasciitis - a Prospective Kohort Study
Brief Title: Proximal Medial Gastriocnemius Recession for Chronic Plantar Fasciitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK317597
Record Dates: First submitted 2021-12-01; First posted 2021-12-17 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Plantar Fasciitis
Keywords: proximal medial gastrocnemius recession; MOxFQ; VAS; EQ5D; MRI; Regression analysis; Ankle movement; Adverse events
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proximal Medial Gastrocnemius Recession Surgery (Experimental): All patients included in the Cohort Study will recieve this PMGR-surgery
  Interventions: Procedure: Proximal Medial Gastrocnemius Recession

INTERVENTIONS:
Procedure: Proximal Medial Gastrocnemius Recession — Patients will be operated with PMGR as described by Barouk. No additional procedures will be performed. The surgery will be performed with the patients in a prone position under local anaesthetics. A 3-4 cm transverse skin incision is made in the popliteal fossa, the superficial fascia is opened, and the medial gastrocnemius with its tendon (aponeurosis) is located. The tendon is then cut while lifting it with clamps, and care is taken to cut only the white tendon while sparing the underlying muscle. While performing a dorsiflexion movement of the ankle, careful palpation of the muscle is done to ensure that all tendon strands are cut completely. The incision is closed in layers, and only soft dressings applied. Patients will be instructed to continue the stretching exercises and fully weight-bear from the first postoperative day. If needed, the patients will be allowed to use crutches during the first 2 weeks after surgery. Sutures are removed 2-3 weeks after surgery.
  Other Names: PMGR

SUMMARY:
This prospective kohort study will follow 150 patients treated with proximal medial gastrocnemius recession for plantar fasciitts. Follow up time is two years and the main outcome is the Manchester Oxford Foot Questionnaire.

A regression analasys will be performed to identify possible patient baseline factors that may affect the effect of surgery,

DETAILED DESCRIPTION:
Recent studies indicate that chronic plantar fasciitis can be treated effectively with Proximal Medial Gastrocnemius Recession (PMGR). In our hospital this treatment has been inocorporated into routine care. This prospective kohort study will follow 150 patients with chronic planatar fasciitis operated with PMGR study. The follow up time is 2 years and the study aims at documenting the effect of the surgery with PROMS (patient related outcome measures), MRI (magnetic resonnance imaging) and ankle movement measurements. 26 patient-related baseline factors will also be registered. A regression analysis will be performed to identify factors that may be predictive to the effect of PMGR surgery.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-75 years.
2. Diagnosis plantar fasciitis verified clinically by orthopaedic surgeon.
3. Diagnosis verified by MRI. MRI criteria: Thickening of the plantar fascia, oedema in the calcaneus, pathological singal changes in the plantar fascia (37)
4. Duration of symptoms must be at least 12 months.
5. An isolated gastrocnemius contracture must be verified with the Silverskiölds test before inclusion.
6. Conventional Physical Therapy must have been tried at least three months without positive effects on symptoms from affected foot.

Exclusion criteria:

1. Previously undergone surgery for plantar fasciitis.
2. Patients with severe talocrural pathology or serious malalignment of foot and ankle
3. Severely reduced peripheral circulation or chronic ulcerations of the foot
4. History of alcoholism, drug abuse, psychological or other emotional problems likely to jeopardize informed consent.
5. Patients with a contraindication/non-compliance for MRI examination.
6. Unable to walk without aid.
7. Not able to read and/or speak a Scandinavian language or English adequately.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Manchester Oxford Foot Questionnaire (MOxFQ) | Baseline
  Patient Related Outcome Measure (PROM) validated for disorders in foot and ankle
Manchester Oxford Foot Questionnaire (MOxFQ) | 6 weeks postoperatively
  Patient Related Outcome Measure (PROM) validated for disorders in foot and ankle
Manchester Oxford Foot Questionnaire (MOxFQ) | 12 weeks postoperatively
  Patient Related Outcome Measure (PROM) validated for disorders in foot and ankle
Manchester Oxford Foot Questionnaire (MOxFQ) | 1 year postoperatively
  Patient Related Outcome Measure (PROM) validated for disorders in foot and ankle
Manchester Oxford Foot Questionnaire (MOxFQ) | 2 years postoperatively
  Patient Related Outcome Measure (PROM) validated for disorders in foot and ankle

SECONDARY OUTCOMES:
VAS (visual analogue scale) | Baseline, 12 weeks, 1 year, 2 years
  Visual analogue scale for pain during use of affected leg in the last 24 hours. 0 is no pain. 10 is worst pain imaginable.
EQ5D (EuroQol questionnaire ) | Baseline, 12 weeks, 1 year, 2 years
  EQ-5D is a validated generic health-related quality-of-life instrument. It consists of two parts: EQ-5D descriptive part and EQ-5D visual analogue scale. The descriptive part includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with three possible answers ("no problems", "some problems", and "major problems"). EQ5D VAS is a visual analogue scale of self-related overall health, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state
MRI (magnetic resonancd imaging) findings | Baseline, 2years
  Thickness of plantar fascia at insertion, pathological signals in the fascia yes/no more, less or same as before, presence of oedema in the calcaneal bone yes/no.
Adverse events | Baseline, 6 weeks, 12 weeks, 1 year, 2 years
  infection, nerve injury, thrombosis.
Ankle movement | Baseline, 12 weeks, 2 years
  Ankle dorsiflexion measured in degrees, through a validated gonimeter
Gait analysis - Maximal ankle dorsiflexion during stance (degrees) | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
  - Maximal ankle dorsiflexion during stance (degrees)
Gait analysis (Length of stride. Centimeters) | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
Gait analysis Ankle power | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
Gait analysis Cadence (steps/minute) | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
Gait analysis Maximal external rotation of ankle during stance (degrees) | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
  * Maximal ankle dorsiflexion during stance (degrees)
  * Length of stride. Centimeters
  * Cadence (steps/minute)
  * Ankle power
  * Maximal external rotation of ankle during stance (degrees)
  * Knee extension while maximal dorsiflexion of ankle during stance (degrees)
Gait analysis Knee extension while maximal dorsiflexion of ankle during stance (degrees) | Baseline, 3 months
  A sub-group of patients (n= 30) will be offered to be tested in a walking lab, comparing their ankle dorsiflexion during stance pre-and postoperatively. Due to a limited access to this facility, not all patients will be able to perform this test.
Assessment of treatment success -pain | at 2 years
  Likert question: I have pain in the heel pain in the leg that was operated two years ago Answers. 1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - physical activity | at 2 years
  Likert question:Heel pain prevents me from performing physical acitvity Answers. 1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - daily living | at 2 years
  Likert question:Heel pain prevents me from performing activities of daily living Answers. 1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - other treatments | at 2 years
  Likert question:I have pain and/or discomfort in the calf that was operated two years ago Answers. 1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - patient acceptable symptom state | at 2 years
  I have received other treatments for plantar fasciitis since surgery was performed two years ago YES/NO
Assessment of treatment success | at 2 years
  If you were to continue having the same level of symptoms in the next few months, would you consider that acceptable.
  YES/NO

OTHER OUTCOMES:
Baseline Patient related factors | Baseline
  The baseline assessment of outcomes and baseline data will be performed no less than two-four weeks before intervention.
  Baseline data includes Age, sex, BMI, smoking, medication, diabetes, rheumatologic disease, employment, type of employment, education level, duration of symptoms, previous treatments, activity level, clinical varus/valgus deformity, use of insoles, previous surgeries in affected foot/ankle for other conditions, clinical hallux valgus deformity, symptomatic hallux valgus deformity, taylors bunion, stable/unstable ankle joint, dominant foot, MRI findings (2), X-ray finding (1): Heel spur. Total number of variables: 26 These data will later be used in regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No